CLINICAL TRIAL: NCT02215005
Title: Steady State Pharmacokinetics of 80 mg Telmisartan (Micardis®), 10 mg Ramipril (Delix®) or the Combination Following Repeated Oral Doses to Healthy Male and Female Volunteers (an Open-label, Randomised, Multiple-dose, Three-way Crossover Study)
Brief Title: Steady State Pharmacokinetics of Telmisartan, Ramipril or the Combination Following Repeated Oral Doses to Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1236.6
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — Telmisartan; Ramipril

ARMS (3):
- Telmisartan + Ramipril (Experimental): 5 days qd
  Interventions: Drug: Telmisartan; Drug: Ramipril
- Telmisartan (Active Comparator): 5 days qd
  Interventions: Drug: Telmisartan
- Ramipril (Active Comparator): 5 days qd
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Telmisartan
  Other Names: Micardis®
  Arms: Telmisartan; Telmisartan + Ramipril
Drug: Ramipril
  Other Names: Delix®
  Arms: Ramipril; Telmisartan + Ramipril

SUMMARY:
The main objective was to investigate the effect of concurrent dosing of 10 mg ramipril and 80 mg telmisartan on the multiple-dose pharmacokinetics of telmisartan and ramipril. Therefore the relative bioavailability of telmisartan and ramipril given in combination was determined in comparison with either telmisartan or ramipril given alone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females according to the following criteria based upon a complete medical history, including the physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory tests
* Age ≥18 and ≤55 years
* Body mass index (BMI) ≥18.5 and ≤29.9 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial (especially unspecific inducing agents like St.John´s wort (Hypericum perforatum) or inhibitors like cimetidine) or drugs that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration of trial drug or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Alcohol abuse (more than 60 g/day) or inability to stop alcoholic beverages for 24 hours prior to dosing and up to the last sampling time point
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration of trial drug or during the trial)
* Excessive physical activities (within one week prior to administration of trial drug or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for torsade de pointes (e.g., heart failure, hyperkalaemia, hypokalemia, family history of Long QT Syndrome)
* Any history of relevant low blood pressure
* Supine blood pressure at screening of systolic <110 mm Hg and diastolic <60 mm Hg
* History of urticaria
* History of angioneurotic edema
* Hereditary fructose intolerance
* Salt and/or volume depletion

For female subjects:

* Pregnancy or planning to become pregnant during the study or within 1 months of study completion
* Positive pregnancy test
* Not willing or unable to use a reliable method of contraception such as implants, injectables, combined oral contraceptives, sterilisation, intrauterine device, double barrier method, sexual abstinence for at least 1 month, or vasectomised partner as only method of contraception for at least 6 months prior to participation in the trial, during and up to 1 month after completion/termination of the trial
* Chronic use of oral contraception containing ethinyl estradiol as the only method of contraception
* Currently lactating

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2007-06; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss (area under the concentration-time curve in plasma at steady state over a uniform dosing interval τ) | up to 72 hours after last drug administration of each treatment
Cmax,ss (maximum measured concentration in plasma at steady state over a uniform dosing interval τ) | up to 72 hours after last drug administration of each treatment

SECONDARY OUTCOMES:
Concentration of the analytes in plasma | 2, 4, and 12 hours after administration of the first dose of each treatment on day 1
pre-dose concentration of the analytes in plasma immediately before the administration of the next dose | pre-dose up to day 5 of each treatment
tmax,ss (time from last dosing to the maximum concentration of the analytes in plasma at steady state) | up to 72 hours after last drug administration of each treatment
Cmin,ss (minimum concentration of the analytes in plasma at steady state over a uniform dosing interval τ) | up to 72 hours after last drug administration of each treatment
Cpre,ss (pre-dose concentration of the analytes in plasma immediately before the administration of the next dose at steady state) | pre-dose up to day 5 of each treatment
Cavg (average concentration of the analytes in plasma at steady state) | up to 72 hours after last drug administration of each treatment
λz,ss (terminal rate constant in plasma at steady state) | up to 72 hours after last drug administration of each treatment
t1/2, ss (terminal half-life of the analyte in plasma at steady state) | up to 72 hours after last drug administration of each treatment
MRTpo,ss (mean residence time of the analyte in the body at steady state after oral administration) | up to 72 hours after last drug administration of each treatment
CL/F,ss (apparent clearance of the analyte in plasma at steady state after extravascular multiple dose administration) | up to 72 hours after last drug administration of each treatment
Vz/F,ss (apparent volume of distribution of the analyte in plasma at steady state after extravascular multiple dose administration) | up to 72 hours after last drug administration of each treatment
PTF (Peak-Trough Fluctuation) | up to 72 hours after last drug administration of each treatment
AUC0-tz,ss (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 72 hours after last drug administration of each treatment
Number of patients with adverse events | up to day 76
Number of patients with clinically relevant changes in Vital Signs (Blood Pressure, Pulse rate) | up to day 76
Number of patients with clinically relevant changes in 12-lead electrocardiogram | up to day 76
Number of patients with clinically relevant changes in laboratory tests | up to day 76
Assessment of tolerability by the investigator on a 4-point scale | Day 8 of each treatment